CLINICAL TRIAL: NCT06147934
Title: Liver and Spleen Stiffness Measured by 2D-shear Wave Elastography for Diagnosis of Liver Fibrosis in Patients With Compensated Advanced Chronic Liver Disease: a Diagnostic Accuracy Study
Brief Title: Liver and Spleen Stiffness Measured by 2D-SWE for Diagnosis of Liver Fibrosis in Patients With cACLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: ZDWY.GRBK.035
Record Dates: First submitted 2023-11-15; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Liver Fibrosis; Liver Cirrhosis
Keywords: 2D-SWE; Liver Cirrhosis; Liver Fibrosis; Liver Stiffness; Spleen Stiffness
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: All participants included will be in one study group.
  Interventions: Diagnostic Test: Diagnostic Test: Transient elastography (TE) and 2D-shear wave elastography (2D-SWE)

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Transient elastography (TE) and 2D-shear wave elastography (2D-SWE) — Index test: TE examination will be completed by experienced nurses, requiring fasting for more than 4 hours before the examination and an interval of no more than 1 week from the abdominal ultrasound and 2D-SWE examination. The report will be considered highly reliable only if IQR/med is ≤ 30%, at least 10 successful acquisitions are obtained, and the success rate is at least 60%. Abdominal ultrasound and 2D-shear wave elastography (2D-SWE) will be completed by a sonographer, the interval between ultrasonic examination and laboratory tests should be less than a week, and the patients should fast for at least 4 hours before the examination.
  Reference standard: Liver biopsy will be conducted by experienced interventionists and reported by pathologists. There should be a maximum interval of no more than 1 month between the liver biopsy and ultrasound examination, and the length of specimen should be more than 1.0cm.

SUMMARY:
A observational diagnostic study will be conducted to evaluate the performance of liver stiffness and spleen stiffness measured by 2D-shear wave elastography (2D-SWE) for diagnosing liver fibrosis in people with compensated Advanced Chronic Liver Disease (cACLD), and explore the cut-off value of 2D-SWE for diagnosing liver fibrosis.

DETAILED DESCRIPTION:
Patients with chronic liver disease who visit Fifth Affiliated Hospital, Sun Yat-Sen University will be enrolled from October 2023 to January 2025. Their liver stiffness measured by transient elastography (TE) should be at least 10 kilopascal (kPa) and with no previous decompensation symptoms.

Patients will be asked to sign an informed consent form. After that, researchers will assess the eligibility of the participants according to inclusion and exclusion criteria, and record their demographic data, history of disease, and the etiology of liver disease.

The participants will be required to complete relevant laboratory tests such as blood routine, liver function, kidney function, coagulation function and etiology. After completing the tests, the results will be recorded by primary researchers.

Abdominal ultrasound and 2D-shear wave elastography (2D-SWE) will be conducted by a sonographer, the interval between ultrasonic examination and laboratory tests should be less than a week, and the patients should fast for at least 4 hours before the examination. Abdominal ultrasound findings, liver stiffness, spleen stiffness, spleen thickness, spleen diameter, portal vein trunk diameter will be recorded by primary researchers.

TE examination will be conducted by experienced nurses, instructing patients to have a fasting period of at least 4 hours prior to the tests. An interval of no more than 1 week should separate the abdominal ultrasound and 2D-SWE examination. The report will be considered highly reliable only if the interquartile range to median ratio (IQR/med) is ≤ 30%, at least 10 successful acquisitions are obtained, and the success rate is at least 60%. Liver stiffness, spleen stiffness and controlled attenuation parameter (CAP) will be recorded by primary researchers.

Liver biopsy will be conducted by experienced interventionists and reported by pathologists. There should be a maximum interval of no more than 1 month between the liver biopsy and ultrasound examination, and the length of specimen should be more than 1.0cm. Primary researchers will record the length of specimen, histological stage, etiology of liver disease, immunohistochemistry results and so on.

Demographic characteristics and laboratory results will be collected to describe participants' condition, and the sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and area under the receiver operating characteristic (AUROC) of 2D-SWE will be compared with that of TE in diagnosing liver fibrosis, and the cut-off value of 2D-SWE for diagnosing liver fibrosis will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years old;
* Chronic liver disease (alcoholic liver disease, chronic hepatitis B, chronic hepatitis C or non-alcoholic fatty liver disease);
* No previous decompensation-related manifestations (such as ascites, gastrointestinal varicose bleeding, hepatic encephalopathy, etc.);
* Informed consent has been signed.

Exclusion Criteria:

* Hepatocellular carcinoma or other advanced malignant tumor;
* Acute liver disease or ALT≥5×ULN;
* Persistent substance abuse other than alcohol;
* Pregnancy or HIV infection;
* There are contraindications of percutaneous liver biopsy (such as serious abnormality of coagulation function, etc.);
* There are conditions that seriously affect TE and 2D-SWE measurements (such as the intercostal space is too narrow, BMI≥30, etc.);
* Subjects considered unsuitable for including in this study but not included by the above exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease who visit Fifth Affiliated Hospital, Sun Yat-Sen University will be enrolled from October 2023 to January 2025. Their liver stiffness measured by transient elastography (TE) should be at least 10kPa no previous decompensation symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 2D-SWE | Through study completion, an average of 2 year
  True Positive/ (True Positive+False Negative) ×100%
Specificity of 2D-SWE | Through study completion, an average of 2 year
  True Negative/ (True Negative+False Positive) ×100%
Positive Predictive Value of 2D-SWE | Through study completion, an average of 2 year
  True Positive/ (True Positive+False Positive) ×100%
Negative Predictive Value of TE and 2D-SWE | Through study completion, an average of 2 year
  True Negative/ (True Negative+False Negative) ×100%
Overall diagnostic performance of TE and 2D-SWE | Through study completion, an average of 2 year
  Measured by the area under the receiver operating characteristic curve (AUROC). The test accuracy level is considered high when the AUROC value is ≥ 0.9.

CONTACTS AND LOCATIONS:
Overall Officials: Xi Liu, PhD, Principal Investigator — The Fifth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- The Fifth Affiliated Hospital, Sun Yat-sen University, Zhuhai, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study will be available from the principal investigator on reasonable request.